CLINICAL TRIAL: NCT06754852
Title: A Phase 1/2 Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of HMB-002 in Participants With Von Willebrand Disease (Velora Pioneer)
Brief Title: A Study Assessing HMB-002 in Participants With Von Willebrand Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hemab ApS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HMB-002-102
Record Dates: First submitted 2024-12-19; First posted 2025-01-01 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Von Willebrand Disease (VWD); Von Willebrand Disease (VWD), Type 1; Von Willebrand Disease (VWD), Type 2
Keywords: Von Willebrand Disease (VMD); Type 1 VWD; Type 2 VWD; Von Willebrand Factor (VWF)
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A Single Ascending Dose Design (Experimental): A multicenter study to evaluate the safety, tolerability, PK, and PD effect of single dose HMB-002 in participants with Type 1 VWD.
  Interventions: Drug: HMB-002 (Part A)
- Part B Multiple Dose Assessment (Experimental): A multicenter study to evaluate the safety, tolerability, PK, and PD effect of 3 repeat doses of HMB-002, as well as the preliminary prophylactic effects on bleeding events.
  Interventions: Drug: HMB-002 (Part B)

INTERVENTIONS:
Drug: HMB-002 (Part A) — HMB-002 will be administered subcutaneously. Part A will utilize sentinel dosing. The planned duration of study participants in Part A is approximately 12 weeks.
  Arms: Part A Single Ascending Dose Design
Drug: HMB-002 (Part B) — HMB-002 will be administered subcutaneously. Part B dosing intervals will be determined following evaluation of Part A results. The planned duration of study participants in Part B will be approximately 21 weeks.
  Arms: Part B Multiple Dose Assessment

SUMMARY:
This is a first-in-human (FIH), Phase 1/2, open-label, dose escalation, safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD), and efficacy study of HMB-002 in participants with VWD. Part A of the study involves a single ascending dose (SAD) design to establish safety, tolerability, PK, and PD effect. In Part B of the study, the safety and tolerability of repeat dosing will be established prior to cohort expansion to explore efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Has the ability to provide informed consent to participate in the study, in accordance with applicable regulations.
2. Has an understanding, ability, and willingness to comply with study procedures and restrictions.
3. ≥18 and <65 years.
4. Weight 50 to 110 kg, inclusive.
5. Congenital Type 1 VWD, Type 1C and Type 2A VWD diagnosis as documented by laboratory results for VWF antigen and activity.
6. Vital signs are within the following ranges at Screening:

   1. Resting pulse rate ≤105 bpm
   2. Blood pressure (BP):

      * Systolic blood pressure: 90 - 140 mmHg
      * Diastolic blood pressure: 40 - 90 mmHg
7. Participants assigned female at birth and of child-bearing potential must have a negative serum pregnancy test within 72 hours prior to the first dose of HMB-002.
8. Women of childbearing potential (CBP) must agree to use two medically acceptable methods of contraception throughout the study. Men with sexual partners of CBP must agree to use a condom please one additional method of contraception (used by their female partner) throughout the study.
9. Participants must meet the following baseline organ function, indicated by laboratory criteria as Screening:

   1. Renal: Estimated glomerular filtration rate (eGFR) of ≥45 ml/min/1.73m^2.
   2. Hepatic: Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and total bilirubin ≤1.5 upper limit of normal (ULN) range at Screening. For participants with a history of Gilbert's Syndrome, total bilirubin ≤2 × ULN.
   3. Hematology (Hgb): Hemoglobin >85 g/L and platelet count >120 x 10^9/L.
10. PART B ONLY- Participants must be symptomatic (typically reporting bleeding events every month) with a minimum of 3 treated bleeding events reported in either the observational study HMB-002-101_SCR or in the participant's medical record.
11. Part B only: Participants may be enrolled if they have completed Part A follow-up.

Exclusion Criteria:

1. History of clinically significant hypersensitivity associated with monoclonal antibody therapies.
2. Personal history of venous or arterial thrombosis or thromboembolic disease, except for catheter-associated, superficial venous thrombosis.
3. High risk thrombophilia: Homozygous Factor V Leiden (FVL), compound heterozygous FVL/Prothrombin gene mutation, Antithrombin <50%. Congenital Protein C and Protein S deficiency with levels <50%.
4. Requires ongoing hemostatic treatment to prevent bleeding, except prior to procedures/surgery.
5. Has a positive test for Hepatitis B surface antigen (HbsAg), Hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at Screening with RNA level above the lower limit of detection.
6. Has received any live vaccine within 28 days prior to signing of informed consent and/or is planning to have a live vaccine during the study period.
7. Planned major surgery during the course of the study.
8. Body mass index (BMI) >35 kg/m^2 (obese, adjusted for ethnicity).
9. Other conditions that substantially increase risk of thrombosis either individually or in combination by the discretion of the Investigator.
10. Participants who are pregnant or breastfeeding.
11. Clinically significant cardiovascular disease.
12. Participants who are currently smoking and unable to refrain from cigarette/cigar/tobacco/vape smoking throughout the study duration.
13. Other conditions that substantially increase the risk of cardiovascular events by the discretion of the Investigator.
14. Congenital or acquired bleeding disorders other than Type 1, Type 1C, or Type 2A VWD.
15. Concurrent disease, treatment, medication (including but not limited to drugs that would affect hemostasis), or abnormality in clinical laboratory tests may pose additional risk in the opinion of the investigator.
16. Hypersensitivity to study drug or any of the excipients.
17. Received investigational medication in another clinical study within 5 half-lives before administration of HMB-002.
18. Requires the use of drugs that would affect hemostasis (including, but not limited to anticoagulation, antiplatelet agents, certain non-steroidal anti-inflammatory drugs) and cannot refrain from use for 14 days prior to the first dose of study drug and throughout the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment emergent adverse events (TEAE) | up to Day 113

SECONDARY OUTCOMES:
Pharmacokinetic Parameter: Maximum observed plasma concentration (Cmax) | Day 1 to Day 113
Pharmacokinetic Parameter: Area under the curve from time zero to last quantifiable concentration (AUClast) | Day 1 to Day 113
Pharmacokinetic Parameter: Area under the curve from time zero to extrapolated infinite time (AUCinf) | Day 1 to Day 113
Pharmacokinetic Parameter: Time to reach maximum observed plasma concentration (Tmax) | Day 1 to Day 113
Pharmacodynamics Parameters: Assessment of VWF antigen (VWF:Ag) | Day 1 to Day 113
Pharmacodynamics Parameters: Assessment of VWF activity | Day 1 to Day 113
Pharmacodynamics Parameters: Assessment of FVIII activity | Day 1 to Day 113
Annualized Bleeding Rate Assessments | Day 1 to Day 113

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (3):
  - Fiona Stanley Hospital, Murdoch, Perth
  - Royal Prince Alfred Hospital, Camperdown, Sydney
  - The Alfred Hospital, Melbourne, Victoria
- Richmond Pharmacology, London, United Kingdom